CLINICAL TRIAL: NCT04110340
Title: An Open-label, Randomised, Non-inferiority Trial of the Efficacy and Safety of Ciprofloxacin Versus an Aminoglycoside Followed by Ciprofloxacin in the Treatment of Bubonic Plague
Brief Title: Ciprofloxacin Versus an Aminoglycoside Followed by Ciprofloxacin for Bubonic Plague
Acronym: IMASOY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Hôpital Universitaire Joseph Raseta Befelatanana CHU d'Antananarivo (Unknown); Institut Pasteur de Madagascar (Other); Foreign, Commonwealth and Development Office and Wellcome (216273.Z.19.Z) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45-18
Record Dates: First submitted 2019-01-28; First posted 2019-10-01 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Plague, Bubonic; Plague, Pneumonic
MeSH Terms: conditions — Plague | interventions — Ciprofloxacin; Streptomycin; Gentamicins

STUDY DESIGN:
Intervention Model Description: An open label, randomised, non-inferiority trial of the efficacy and safety of ciprofloxacin versus an aminoglycoside + ciprofloxacin in treatment of bubonic plague. We are using a non-inferiority design since the overall cure rate for bubonic plague without septicaemia with streptomycin is approximately 95%. As a result, demonstrating superiority would be unnecessary and impractical given the sample size that would be required. Our aim is therefore to demonstrate that ciprofloxacin alone is not more than 15% inferior to an aminoglycoside followed by ciprofloxacin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofloxacin Arm (Active Comparator): Adults: Ciprofloxacin 500mg orally twice daily (or 400mg IV twice daily for those who cannot take oral medication) for 10 days;
  Children:Ciprofloxacin 15mg/kg twice daily (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take oral - maximum dose 400mg) for 10 days.
  Interventions: Drug: Ciprofloxacin
- Control arm (Other): Adults: streptomycin 1g twice daily for three days, followed by ciprofloxacin 500mg orally twice daily (or ciprofloxacin 400mg twice daily by IV for those who cannot take it orally) for an additional 7 days.
  OR
  2.5mg/kg IV gentamicin twice daily for 3 days followed by ciprofloxacin 500 mg orally twice daily (or ciprofloxacin 400 mg twice daily IV for those who cannot take oral) for a further 7 days.
  Children: streptomycin 15mg/kg twice daily for three days followed by ciprofloxacin 15mg/kg twice daily (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take oral - maximum dose 400mg) for 7 additional days.
  OR
  2.5mg/kg IV gentamicin twice daily for 3 days, followed by ciprofloxacin 15mg/kg (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take the oral route) for a further 7 days.
  Interventions: Drug: Ciprofloxacin; Drug: Streptomycin; Drug: Gentamicin

INTERVENTIONS:
Drug: Ciprofloxacin — Adults: Ciprofloxacin 500mg orally twice daily (or 400mg IV twice daily for those who cannot take oral medication) for 10 days;
  Children:Ciprofloxacin 15mg/kg twice daily (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take oral - maximum dose 400mg) for 10 days.
  Patients who begin intravenous therapy may switch to oral administration once they are able to swallow or once deemed clinically appropriate by the treating physician.
Drug: Streptomycin — Adults: streptomycin 1g twice daily for three days, followed by ciprofloxacin 500mg orally twice daily (or ciprofloxacin 400mg twice daily by IV for those unable to take orally) for an additional 7 days.
  Children: streptomycin 15mg/kg twice daily for three days followed by ciprofloxacin 15mg/kg twice daily (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take oral - maximum dose 400mg) for 7 additional days.
  Patients who begin intravenous therapy may switch to oral administration once they are able to swallow or once deemed clinically appropriate by the treating physician.
  Arms: Control arm
Drug: Gentamicin — Adults: 2.5mg/kg IV gentamicin twice daily for 3 days followed by ciprofloxacin 500 mg orally twice daily (or ciprofloxacin 400 mg twice daily IV for those who cannot take oral) for a further 7 days.
  Children: 2.5mg/kg IV gentamicin twice daily for 3 days, followed by ciprofloxacin 15mg/kg (max 500mg per dose) orally (or 10mg/kg IV twice daily for those who cannot take the oral route) for a further 7 days.
  Arms: Control arm

SUMMARY:
The primary objective of this trial is to test the hypothesis that ciprofloxacin monotherapy given (orally, intravenously, or combination) for 10 days is non-inferior to an aminoglycoside (given on days 1-3) followed by ciprofloxacin (given on days 4-10) in the treatment of bubonic plague.

Secondary objectives are:

- to evaluate the level and kinetics of anti-Y. pestis antibodies of patients (bubonic and pneumonic plague) included in the study (anti-F1 ELISA techniques) at D1, D11, D21, M3 for patients who are positive at D21, and M12 for patients who are positive at M3.

The tertiary objectives are:

- to evaluate the level and kinetics of the levels of anti-Y. pestis antibodies and circulating F1 antigen of the patients (bubonic and pneumonic plague) included in the study (Luminex MagPix techniques with a Multiplex containing anti-F1 and rLcrV antigens and an F1 antigen capture multiplex) at D1, D11, D21, M3 for patients positive at D21, and M12 for patients who are positive at M3.

Observational non-comparative study of pneumonic plague

* The primary objective is to document the efficacy and safety of the currently recommended combination therapy treatment of pneumonic plague - an aminoglycoside (streptomycin or gentamicin) and ciprofloxacin combination therapy.
* The secondary and tertiary objectives of the bubonic plague trial also apply to the pneumonic plague cohort.

DETAILED DESCRIPTION:
An individually randomised, open label, non-inferiority trial of ciprofloxacin versus an aminoglycoside and ciprofloxacin in patients with bubonic plague. We are using a non-inferiority design since the overall cure rate for bubonic plague without septicaemia with streptomycin is approximately 95%. As a result, demonstrating superiority would be unnecessary and impractical given the sample size that would be required. Our aim is therefore to demonstrate that ciprofloxacin alone is not more than 15% inferior to an aminoglycoside followed by ciprofloxacin. (15% is the non-inferiority margin in our study). We will recruit patients with a clinical suspicion of bubonic plague, but the size of our sample is powered based on an intention to treat infected patients sample size of 190, where infected is defined as a confirmed or probable case of bubonic plague. As a result the total number of patients to be enrolled will be higher than 190. We estimate that we will need to recruit approximately 600 patients with bubonic plague to achieve a sample size of 190 confirmed/probable bubonic plague patients. However, to mitigate risks of being under-powered we will propose to recruit for three full seasons with a minimum target of 190 confirmed/probable cases. Should we achieve the target of 190 confirmed/probable bubonic plague cases before the end of the final transmission season, we will nevertheless continue to recruit until the end of the season to retain power in the event of different treatment success percentages and to allow us to increase precision.

We will also recruit and collect data on patients with pneumonic plague, who will be enrolled in to a parallel observational cohort.

ELIGIBILITY:
Inclusion Criteria for randomisation to the bubonic plague treatment trial:

Bubonic plague

* Patients of any age AND
* Recent onset (< 10 days) of fever (uncorrected axillary temperature ≥ 37.5C) or history of fever AND
* One or more buboes (tender lymph node swelling) AND
* Residence or travel to a plague endemic area in Madagascar within 14 days of the onset of symptoms AND
* Patients identified as clinically suspected of plague by health personnel (doctors or paramedics)

Exclusion Criteria to the bubonic plague treatment trial:

* Known allergy to aminoglycosides or fluoroquinolones
* Tendinitis
* Myasthenia gravis
* Theophylline or warfarin use
* Already treated for bubonic or pneumonic plague in the preceeding 3 months
* Women who report being pregnant

Inclusion of patients to the pneumonic plague observational cohort:

• Suspected, probable and confirmed cases of pneumonic plague

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with bubonic plague with a therapeutic response (assessed on day 11).Therapeutic response is defined as follows for subjects with a visible bubo: | 11 days
  * Alive
  * Absence of fever
  * Has not received alternative treatment for plague
  * No clinical decision to continue anti-plague antibiotics beyond day 10

SECONDARY OUTCOMES:
Bubonic plague | 4 days
  • Proportion of patients without fever (uncorrected axillary temperature <37.5C) at Day 4
Bubonic plague | 4 days
  • Proportion of patients with a pain score < 3 at Day 4 (using pain scale questionnaires)
Bubonic plague | 11 days
  • Proportion of patients with a pain score < 3 at Day 11 (using pain scale questionnaires)
Bubonic plague | 4 days
  • Mean % change in bubo size at Day 4 (measured by use of calipers and/or ultrasound)
Bubonic plague | 11 days
  • Mean % change in bubo size at Day11 (measured by use of calipers and/or ultrasound)
Bubonic plague | 4 days
  • Proportion of patients experiencing a serious adverse event on or before Day 4
Bubonic plague | 11 days
  • Proportion of patients experiencing a serious adverse event on or before Day 11
Bubonic plague | 21 days
  • Proportion of patients experiencing a serious adverse event on or before Day 21
Bubonic plague | 21 days
  • Proportion of patients who are fully adherent to the study treatment schedule.
Pneumonic plague | 11 days
  Proportion of patients with a therapeutic response at Day 11. Therapeutic response is defined as follows:
  * Alive
  * Resolution of fever (uncorrected axillary temperature <37.5C)
  * Resolution of tachypnoea (RR< 24 in adults, but age-specific in children)
Pneumonic plague | 4 days
  • Proportion of patients without fever (uncorrected axillary temperature <37.5C) at Day 4
Pneumonic plague | 4 days
  • Proportion of patients with tachypnoea resolution (RR< 24 in adults, but age-specific in children) at Day 4
Pneumonic plague | 4 days
  • Proportion of patients experiencing a serious adverse event on or before Day 4
Pneumonic plague | 11 days
  • Proportion of patients experiencing a serious adverse event on or before Day 11
Pneumonic plague | 21 days
  • Proportion of patients experiencing a serious adverse event on or before Day 21
Pneumonic plague | 21 days
  • Proportion of patients who are fully adherent to the study treatment schedule.
Therapeutic response is defined as follows for subjects with a visible bubo: | 11 days
  * Alive AND
  * Absence of fever at D11 AND
  * At least a 25% decrease in bubo size (in the case of multiple buboes, the largest bubo) AND
  * Has not received alternative treatment for plague AND
  * No clinical decision to continue anti-plague antibiotics beyond day 10
    ● Therapeutic response is defined as follows for subjects with small buboes that are palpable but not measurable:
  * Alive AND
  * Absence of fever at D11 AND
  * Bubo has not enlarged AND
  * Has not received alternative treatment for plague AND
  * No clinical decision to continue anti-plague antibiotics beyond day 10

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Horby, MD, Principal Investigator — University of Oxford
Locations (1):
- Professor Mamy Randria, Antananarivo, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data relating to the published analyses will be made available through an existing online repository (either at the University of Oxford or LSHTM) once the trial results are published.
Time Frame: Anticipated release date: May 2025
Access Criteria: To be confirmed

REFERENCES:
- [Derived] Randremanana RV, Raberahona M, Bourner J, Rajerison M, Edwards T, Randriamparany R, Fehizoro Razafindratsinana T, Razananaivo LH, Zadonirina G, Mayouya-Gamana T, Salam APA, Mangahasimbola RT, Andrianaivoarimanana V, Pesonel E, Rakotoarivelo RA, Randria MJD, Horby P, Olliaro P; IMASOY Study Group. Ciprofloxacin versus Aminoglycoside-Ciprofloxacin for Bubonic Plague. N Engl J Med. 2025 Aug 7;393(6):544-555. doi: 10.1056/NEJMoa2413772. PMID 40768716
- [Derived] Randremanana RV, Raberahona M, de Dieu Randria MJ, Bourner J, Zadonirina G, Razananaivo H, Mayouya-Gamana T, Mangahasimbola R, Pesonel E, Gillesen A, Rajerison M, Andrianaivoarimanana V, Edwards T, Horby P, Olliaro P. An open-label, randomized, non-inferiority trial of the efficacy and safety of ciprofloxacin versus an aminoglycoside + ciprofloxacin in the treatment of bubonic plague (IMASOY): study protocol for a randomized control trial-an update to the published protocol. Trials. 2024 Jul 5;25(1):457. doi: 10.1186/s13063-024-08302-7. PMID 38970065
- [Derived] Randremanana RV, Raberahona M, Randria MJD, Rajerison M, Andrianaivoarimanana V, Legrand A, Rasoanaivo TF, Randriamparany R, Mayouya-Gamana T, Mangahasimbola R, Bourner J, Salam A, Gillesen A, Edwards T, Schoenhals M, Baril L, Horby P, Olliaro P. An open-label, randomized, non-inferiority trial of the efficacy and safety of ciprofloxacin versus streptomycin + ciprofloxacin in the treatment of bubonic plague (IMASOY): study protocol for a randomized control trial. Trials. 2020 Aug 17;21(1):722. doi: 10.1186/s13063-020-04642-2. PMID 32807214